CLINICAL TRIAL: NCT01559649
Title: Development and Validation of a VA Stroke Swallowing Screening Tool
Brief Title: Stroke Swallowing Screening Tool Validation
Acronym: SSST
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C7242-R
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Results first posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-06

CONDITIONS: Cerebrovascular Disorders; Deglutition Disorders
Keywords: Stroke; Deglutition; Deglutition Disorders; Nurse Screening
MeSH Terms: conditions — Cerebrovascular Disorders; Deglutition Disorders; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — no samples will be collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Veterans admitted to MEDVAMC with a suspected ischemic or hemorrhagic stroke will be recruited. Individuals with a history of neurological disease other than stroke, head and neck structural surgery, or history of dysphagia unrelated to the current stroke will be excluded from participation. Individuals who are obtunded, medically unstable, greater than 5 days post-admission will be excluded. Patients with language or cognitive deficits who are judged by the attending neurologist to not have capacity to provide informed consent will be eligible to participate, but they must have an authorized representative available within 24 hours of admission to provide consent. Patients will undergo swallowing screening and videofluoroscopic swallowing study to establish validity of screening items
  Interventions: Behavioral: Establishing Validity and Reliability
- Group 2: Stroke ward nurses. The nurses will administer and interpret the swallowing screening items. Speech pathologists will also make blinded, simultaneous interpretations of the screening items. Nurse and speech pathologist interpretation will be used to establish nursing reliability.
  Interventions: Behavioral: Establishing Validity and Reliability

INTERVENTIONS:
Behavioral: Establishing Validity and Reliability — Consecutive individuals admitted with suspected stroke will be recruited to participate. Individuals will undergo screening of swallowing and a videofluoroscopic swallow study within two hours. Eight screening items will be tested for validity and inter-rater reliability: 6 nonswallowing features and 2 swallowing features. Reliability in nursing observations of each screening item will be completed in all participants. Speech pathologists trained in the screening items will serve as the reference standard from which to compare reliability with registered nurses who routinely work on the hospital ward with stroke patients

SUMMARY:
Stroke is a major medical problem in the United States, and veterans are at significant risk given that the most critical risk factors of stroke, older age and associated medical problems such as high blood pressure, are common. Dysphagia, swallowing problems, can lead to aspiration which in turn may result increased pneumonia, particularly in stroke patients. Development and implementation of an accurate and consistent nursing swallowing screening tool to identify risk of aspiration in individuals admitted with suspected stroke is critical as it allows for immediate intervention, thereby reducing associated medical complications, length of stay, and healthcare costs. The availability of such screening tools, however, is limited. The primary objective of this study is to construct a reliable and valid swallowing screening tool to identify risk of aspiration in individuals admitted with suspected stroke.

DETAILED DESCRIPTION:
Early detection of aspiration risk in acute stroke is critical as it allows for immediate intervention, thereby reducing mortality, morbidity, length of hospitalization, and healthcare costs. Screening of swallowing prior to the administration of food, liquid or medication, including aspirin, in individuals presenting with stroke symptoms is a guideline American Heart Association/American Stroke Association. In accordance with this guideline, the Veterans Health Administration (VHA) has advocated the screening of swallowing be a quality performance measure in acute stroke. Moreover, the Office of the Inspector General recently issued VHA Directive 2006-032 mandating that the initial nurse assessment must include a screening of swallowing. In response to the directive, many VHA facilities created and implemented some version of a nursing swallowing screening tool (SST), but to our knowledge, none have been validated using an instrumental swallowing examination nor has reliability been established. In developing and establishing a valid and reproducible SST for patients with stroke, clinicians are divided on the need to include trial water swallows as part of the SST. The current notion is that administering trial swallows by disciplines without expertise in dysphagia would compromise patient safety, thus this step is opposed by many speech pathologists and nurses. The prudency of introducing non-validated, non-reproducible SSTs is questionable. The primary objective of this study is to construct a reliable and valid SST to identify risk of aspiration in individuals admitted with suspected stroke. The specific aims of this proposal are to: 1) determine if nurses can make reliable inter-rater judgments of swallowing and non-swallowing features historically used by speech pathologists to make judgments of aspiration, and 2) identify the combination of items that provide the highest level of both sensitivity and specificity in the identification of aspiration risk as measured by a videofluoroscopic swallow study (VFSS) in individuals admitted with suspected stroke. Outcomes of this research will inform as to the execution of a multi-site feasibility study on the implementation of a reliable and valid SST by nurses Methods: Consecutive individuals admitted with suspected stroke (N = 270) will be recruited to participate. Individuals will undergo screening of swallowing and a VFSS. Screening items selected for validation in the identification of risk of aspiration in patients presenting with stroke symptoms were based on extensive literature review using Cochrane and QUADAS guidelines. Eight screening items will be tested for validity and inter-rater reliability: 6 non-swallowing features and 2 swallowing features. Reliability in nursing observations of each screening item will be completed in all participants. Speech pathologists will serve as the reference standard from which to compare reliability with registered nurses who routinely work on the hospital ward with stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Veterans of all ethnicities admitted to MEDVAMC with a new suspected ischemic or hemorrhagic stroke will be eligible to participate.
* Individuals with a history of prior strokes without dysphagia will be eligible to participate.
* Patients must be medically stable as determined by the attending neurologist.
* Participants with language or cognitive deficits who are judged by the attending neurologist to not have capacity to provide informed consent will be eligible to participate but they must have an authorized representative available within 24 hours of admission to provide consent.

Exclusion Criteria:

* Individuals with a history of neurological disease other than stroke, head and neck structural surgery, or history of dysphagia unrelated to the current stroke will be excluded from participation.
* Individuals who are obtunded (unable to maintain wakefulness), currently diagnosed with pneumonia, or on ventilator support will be excluded.
* Veterans who are more than 72 hours past MEDVAMC admission will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Veterans admitted with stroke symptoms
  * Nurses working on the stroke ward
Sampling Method: Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2012-10; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie K Daniels, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daniels SK, Pathak S, Stach CB, Mohr TM, Morgan RO, Anderson JA. Speech Pathology Reliability for Stroke Swallowing Screening Items. Dysphagia. 2015 Oct;30(5):565-70. doi: 10.1007/s00455-015-9638-x. Epub 2015 Jul 24. PMID 26205434
- [Result] Daniels SK, Pathak S, Rosenbek JC, Morgan RO, Anderson JA. Rapid Aspiration Screening for Suspected Stroke: Part 1: Development and Validation. Arch Phys Med Rehabil. 2016 Sep;97(9):1440-1448. doi: 10.1016/j.apmr.2016.03.025. Epub 2016 Apr 23. PMID 27117382
- [Result] Anderson JA, Pathak S, Rosenbek JC, Morgan RO, Daniels SK. Rapid Aspiration Screening for Suspected Stroke: Part 2: Initial and Sustained Nurse Accuracy and Reliability. Arch Phys Med Rehabil. 2016 Sep;97(9):1449-1455. doi: 10.1016/j.apmr.2016.03.024. Epub 2016 Apr 24. PMID 27117381
- [Result] Freeland TR, Pathak S, Garrett RR, Anderson JA, Daniels SK. Using Medical Mannequins to Train Nurses in Stroke Swallowing Screening. Dysphagia. 2016 Feb;31(1):104-10. doi: 10.1007/s00455-015-9666-6. Epub 2015 Oct 30. PMID 26519043

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Chart review-1042 suspected stroke patients . Excluded-636 (h/o neuro disease, etc). Eligible-406. 137-declined, d/c before approaching. Consented-269. Screening completed-258 (11-unable to complete screening-d/c, unstable, etc). VFSS completed-256-250 analyzed (6 excluded from analysis-equipment failure, h/o dysphagia, etc.). RNs-15 participated.
Groups:
- Patients With Suspected Stroke: Veterans admitted to MEDVAMC with a suspected ischemic or hemorrhagic stroke recruited. Individuals with a history of neurological disease other than stroke, head and neck structural surgery, or history of dysphagia unrelated to the current stroke were excluded . Individuals who were obtunded, medically unstable, greater than 5 days post-admission were excluded. Patients with language or cognitive deficits who were judged by the attending neurologist to not have capacity to provide informed consent were eligible to participate, but they had to have an authorized representative available within 24 hours of admission to provide consent. Patients underwent swallowing screening and videofluoroscopic swallowing study (VFSS) to establish validity of screening items
- Registered Nurses: Stroke ward nurses. The nurses administered and interpret the swallowing screening items. Speech pathologists made blinded, simultaneous interpretations of the screening items. Nurse and speech pathologist interpretation were used to establish nursing reliability.
Period: Overall Study
Arm/Group | Patients With Suspected Stroke | Registered Nurses
Started | 269 | 15 (Started with 10 nurses. As an RN dropped out due to scheduling, etc, RN replaced with another RN)
Completed | 250 (Screening not completed in 11, VFSS not completed in 2, 6 excluded from analysis. N=250 analyzed) | 9
Not Completed | 19 | 6

BASELINE CHARACTERISTICS:
Population: N=250 stroke patients with data analyzed
Groups:
- Suspected Stroke: Veterans admitted to MEDVAMC with a suspected ischemic or hemorrhagic stroke.
- Nurses: Registered nurses working on MEDVAMC stroke wards
- Total: Total of all reporting groups
Arm/Group | Suspected Stroke | Nurses | Total
Number analyzed (Participants) | 250 | 15 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9.5) | NA (NA) — Age data were not collected for nurses. | NA (NA) — Age data were not collected for nurses.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 243 | 2 | 245
Race/Ethnicity, Customized [Number; unit: participants]
  White | 98 | 1 | 99
  African American | 120 | 3 | 123
  Hispanic | 32 | 5 | 37
  Asian | 0 | 6 | 6
Region of Enrollment [Number; unit: participants]
  United States | 250 | 15 | 265
Previous History of Stroke [Number; unit: participants] | 60 | NA — Number of strokes not collected in nurses. | NA — Total not calculated because data are not available (NA) in one or more arms.
National Institutes of Health Stroke Scale score [Mean (Standard Deviation); unit: units on a scale] — Scores range is 0-30. Lower scores indicates milder stroke.
  units on a scale | 2.6 (2.9) | NA (NA) — Scores not collected for nurses. | NA (NA) — Scores not collected for nurses
Discharge Diagnosis [Number; unit: participants]
  Imaging-confirmed stroke | 140 | NA — discharge diagnosis not collected for nurses | NA — Total not calculated because data are not available (NA) in one or more arms.
  Physician-confirmed stroke | 16 | NA — discharge diagnosis not collected for nurses | NA — Total not calculated because data are not available (NA) in one or more arms.
  Physician-confirmed TIA | 49 | NA — discharge diagnosis not collected for nurses | NA — Total not calculated because data are not available (NA) in one or more arms.
  Nonstroke/TIA | 45 | NA — discharge diagnosis not collected for nurses | NA — Total not calculated because data are not available (NA) in one or more arms.
Stroke Type [Number; unit: participants] — number obtained from the number of imaging confirmed stroke (n=140)
  participants
    Ischemic | 137 | NA — stroke type not collected in nurses | NA — Total not calculated because data are not available (NA) in one or more arms.
    Hemorrhagic | 3 | NA — stroke type not collected in nurses | NA — Total not calculated because data are not available (NA) in one or more arms.
Stroke Location [Number; unit: participants] — obtained from 140 imaging-confirmed strokes
  participants
    right hemispheric damage | 51 | NA — stroke location not collected in nurses | NA — Total not calculated because data are not available (NA) in one or more arms.
    left hemispheric damage | 50 | NA — stroke location not collected in nurses | NA — Total not calculated because data are not available (NA) in one or more arms.
    bilateral | 4 | NA — stroke location not collected in nurses | NA — Total not calculated because data are not available (NA) in one or more arms.
    posterior circulation | 35 | NA — stroke location not collected in nurses | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Screening Items
Description: Identify the combination of screenings items that provide the highest level of sensitivity in the identification of aspiration risk as measured by a videofluoroscopic swallow study (VFSS) in individuals admitted with suspected stroke.
Time Frame: 3 years
Population: Nurses were not assessed for this outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Patients With Suspected Stroke: Veterans admitted to MEDVAMC with a suspected ischemic or hemorrhagic stroke
- Registered Nurses: Stroke ward nurses.
Arm/Group | Patients With Suspected Stroke | Registered Nurses
Number analyzed (Participants) | 250 | 0
percentage of agreement
  Age >70 | 37.9 [20.7 to 57.7] |
  Lethargy | 3.5 [0.087 to 178] |
  Dysarthria | 62.1 [42.3 to 79.3] |
  Nonswallow wet voice | 10.3 [2.19 to 27.4] |
  Abnormal volitional cough | 27.6 [12.7 to 47.2] |
  Combined water swallow items | 72.4 [52.8 to 87.3] |
  Dysarthria or Water swallow item | 86.2 [68.3 to 96.1] |
  Age >70 or Dysarthria or Water swallow item | 93.1 [77.2 to 99.2] |

2. Primary Outcome: Specificity of Screening Items
Description: Identify the combination of screenings items that provide the highest level of specificity in the identification of aspiration risk as measured by a videofluoroscopic swallow study (VFSS) in individuals admitted with suspected stroke.
Time Frame: 3 years
Population: Nurses were not assessed for this outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Arm/Group | Patients With Suspected Stroke | Registered Nurses
Number analyzed (Participants) | 250 | 0
percentage of agreement
  Age >70 | 82.8 [77.2 to 87.5] |
  Lethargy | 99.5 [97.5 to 100] |
  Dysarthria | 80.5 [74.7 to 85.5] |
  Nonswallow wet voice | 98.6 [96.1 to 99.7] |
  Abnormal volitional cough | 95.9 [92.4 to 98.1] |
  Combined water swallow item | 59.7 [52.9 to 66.3] |
  Dysarthria or Water swallow item | 49.3 [42.6 to 56.1] |
  Age >70 or Dysarthria or Water swallow item | 43.0 [36.4 to 49.8] |

3. Primary Outcome: Negative Predictive Value of Screening Items
Description: Identify the combination of screenings items that provide the highest level of negative predictive value in the identification of aspiration risk as measured by a videofluoroscopic swallow study (VFSS) in individuals admitted with suspected stroke.
Time Frame: 3 years
Population: Nurses were not assessed for this outcome measure
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Arm/Group | Patients With Suspected Stroke | Registered Nurses
Number analyzed (Participants) | 250 | 0
percentage of agreement
  Age >70 | 91.0 [86.2 to 94.6] |
  Lethargy | 88.7 [84.1 to 92.4] |
  Dysarthria | 94.2 [89.8 to 97.1] |
  Nonswallow wet voice | 89.3 [84.8 to 92.9] |
  Abnormal volitional cough | 91.0 [86.6 to 94.3] |
  Combined water swallow itmes | 94.3 [89.1 to 97.5] |
  Dysarthria or Water swallow item | 96.5 [91.2 to 99.0] |
  Age >70 or Dysarthria or Water swallow item | 97.9 [92.7 to 99.7] |

4. Secondary Outcome: Average Accuracy Rate for Nurse Administration for All Screening Procedures
Description: Determine if current stroke-ward staff nurses can accurately administer screening items.
Time Frame: 3 years
Measure: Mean (Full Range); unit: percentage of accuracy
Groups:
- Nurses: Only nurses administered and interpreted the screening items.
Arm/Group | Nurses
Number analyzed (Participants) | 15
percentage of accuracy | 98.33 [95.42 to 100]

5. Secondary Outcome: Reliability of Nurse Interpretation of Each Screening Items and the Valid Combination of Items
Description: Determine if stroke-ward staff nurses can make reliable inter-rater judgments of swallowing (e.g. cough after swallow, wet voice after swallow) and nonswallowing features (e.g. decreased volitional cough, dysarthria) historically used by SLPs to make judgments of aspiration.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: kappa
Arm/Group | Nurses
Number analyzed (Participants) | 15
kappa
  Lethargy | 0.394 [-0.152 to 0.940]
  Dysarthria | 0.717 [0.667 to 0.754]
  Abnormal volitional cough | 0.645 [0.594 to 0.712]
  Nonswallow wet voice | 0.360 [-0.017 to 0.594]
  Cough after swallowing | 0.911 [0.824 to 0.997]
  Throat clear after swallowing | 0.837 [0.760 to 0.914]
  Wet voice after swallowing | 0.727 [0.567 to 0.888]
  Inability to continuously drink 90ml of water | 0.911 [0.788 to 1.000]
  1 minute wet voice | 1.000 [1.000 to 1.000]

ADVERSE EVENTS:
Time Frame: 30 days post-discharge
Description: Only suspected stroke patients were monitored for pulmonary complications.
Groups:
- Patients With Suspected Stroke: Individuals admitted with suspected ischemic or hemorrhagic stroke
Arm/Group | Patients With Suspected Stroke
Serious Adverse Events (participants affected / at risk) | 0/250
Other Adverse Events (participants affected / at risk) | 0/250

LIMITATIONS AND CAVEATS:
Large number of individuals excluded from participation due to stringent inclusion/exclusion criteria to ensure that stroke-related aspiration was being measured. Small number of women recruited. Inability to screen in the emergency department.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes